CLINICAL TRIAL: NCT06277414
Title: Machine Learning for the Prediction of Post-Endoscopic Retrograde Cholangiopancreatography Complication Risk
Brief Title: a Prediction of Post-Endoscopic Retrograde Cholangiopancreatography Complication
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor
Other Study IDs: 2024ll0204001
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — The blood will be collected and detected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERCP: The postoperative laboratory test results, imaging results and symptoms were collected
  Interventions: Other: collection of laboratory test results, imaging results and symptoms

INTERVENTIONS:
Other: collection of laboratory test results, imaging results and symptoms — collection of laboratory test results, imaging results and symptoms

SUMMARY:
To develop effective preoperative and postoperative prediction models for postoperative complications of ERCP

DETAILED DESCRIPTION:
To develop effective preoperative and postoperative prediction models for postoperative complications of ERCP based on machine learning

ELIGIBILITY:
Inclusion Criteria:

* Routine ERCP patients

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Pregnant women or breastfeeding
* current acute pancreatitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine ERCP patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Pancreatitis | 1 month
  Typical abdominal pain, with the level of serum amylase increasing at least 3 times of the normal range within 24 hours after ERCP.

SECONDARY OUTCOMES:
Number of Acute PEC(post-ERCP-cholecystitis ) | 1 month
  Number of Acute PEC(post-ERCP-cholecystitis )
Number of Participants with Cholangitis | 1 month
  Temperature should be more than 38 celsius degree, chills, with right upper abdominal pain, blood routine showing the total amount of the White Blood Cell (WBC), and the amount of polymorphonuclear neutrophil(PMN) are above normal
Number of Participants with Perforation | 1 month
  Typical abdominal pain,abdominal muscle tension, and there are also radiographic evidence suggesting
Number of Participants with bile duct stents | 1 month
  If it is necessary to get the patients drainage, Number of Participants with stents or endoscopic nasobiliary drainage (ENBD) should be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided